CLINICAL TRIAL: NCT01151696
Title: Prise en Charge Pharmacologique de l'anxiété et de la Douleur Chez Les Patients Qui Souffrent en Situation d'Urgence Traumatique pré-hospitalière : étude randomisée contrôlée en Double Aveugle
Brief Title: Pain and Anxiety Management of Traumatic Emergency in a Pre-hospital Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0918703; 2009-015529-35 (EudraCT Number)
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Pain
Keywords: Pain; morphine; hydroxyzine; acute pain; traumatic pain; anxiety; post trauma stress; post trauma anxiety; post trauma disorders
MeSH Terms: conditions — Pain; Acute Pain; Anxiety Disorders | interventions — Hydroxyzine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- hydroxyzine (Experimental): Patients will receive intravenous hydroxyzine 1mg/kg at the beginning of the morphine titration protocol, and intravenous morphine 0.15 mg/kg then 0.05 mg/kg if necessary, every 5 minutes.
  Interventions: Drug: Atarax (Hydroxyzine)
- Placebo (Placebo Comparator): Patients will receive intravenous placebo at the beginning of the morphine titration protocol, and intravenous morphine 0.15 mg/kg then 0.05 mg/kg if necessary, every 5 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atarax (Hydroxyzine) — One milligram per 10 kilogram, intramuscular use
  Arms: hydroxyzine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Unexpected acute pain in an emergency setting causes anxiety, insecurity, and stress that can diminish perceptions of control over pain and diminish ability to decrease pain. This may interfere with the opioid treatment and poses the question of whether an anxiolytic drug added to the morphine titration could relief pain and/or anxiety. This randomized double-blind group clinical trial is designed to determine the efficacy and safety of hydroxyzine in addition to a conventional intravenous morphine titration protocol.

DETAILED DESCRIPTION:
Obtaining high-quality analgesia in prehospital patients with severe pain is an important treatment objective for medical team. Opioids are recognized as the treatment of choice for relief of severe acute pain. Recommended initial analgesia of patients with severe acute pain, defined as a numerical rating scale (NRS) score of 6/10 or higher, in a prehospital setting in France consists of the administration of morphine by the medical staff of mobile intensive care units. The intravenous administration of morphine is usually considered as the gold standard for any emergency setting. Nevertheless, even when using high dose boluses and aggressive titration protocols, pain relief remains inconsistent for some patients. Moreover, unexpected acute pain in an emergency setting causes anxiety, insecurity, and stress that can diminish perceptions of control over pain and diminish ability to decrease pain. This may interfere with the opioid treatment and poses the question of whether an anxiolytic drug added to the morphine titration could relief pain and/or anxiety.There is no study, to our knowledge, assessing the clinical efficacy of hydroxyzine added to the morphine in a prehospital setting. Hydroxyzine is used primarily as an antihistamine drug for the treatment of itching, allergies, motion sickness-induced nausea, and insomnia, as well as notably for the treatment of mild anxiety. This randomized double-blind group clinical trial is designed to determine the efficacy and safety of hydroxyzine in addition to a conventional intravenous morphine titration protocol by comparing hydroxyzine and placebo for medical prehospital treatment of adult patients with severe traumatic acute pain. Eligible patients with a numerical rating scale (NRS) score of 6/10 or higher will be randomly allocated to receive either hydroxyzine 1mg/kg at inclusion (group A) or an intravenous placebo. The intravenous morphine analgesia will be given and titrated according to the pain score every 5 minutes. The drugs will be administered by the physician from syringes of similar appearance prepared by the nurse who is not otherwise involved in the study. The protocol-defined primary outcome measure is the percentage of patients with pain relief (with a NRS score of 3/10 or lower) 15 minutes after the first injection. Secondary outcomes include pain score comparisons every 5 minutes within the first 30 minutes and comparison of adverse events. The physician blinded to the analgesic treatment groups will do all assessments of patients. The safety evaluation will include non invasive monitoring of blood pressure, heart rate, respiratory rate, oxygen saturation by pulse oximetry (Spo2), and a sedation scale (0, patient is awake; 1, patient is with intermittent sleeping; 2, patient is sleeping, awakened by verbal stimulation; 3, patient is sleeping, awakened by tactile stimulation; 4, patient is not aroused by stimulation) at these periods. Fifteen minutes after the first injection, overall patient and investigator satisfaction with analgesia will be recorded. Moreover, several assessments will be done by psychologists 2 and 21 days after the trauma, including post traumatic stress and anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patient with a severe traumatic acute pain defined by an NRS score of 6/10 or higher at randomization.

Exclusion Criteria:

* Patient-reported history of chronic respiratory, renal, or hepatic insufficiency
* Patient known opioid or hydroxyzine allergies
* recent treatment with opioids or anxiolytics
* incapacity to understand the NRS
* hypotension (defined as a systolic blood pressure <90 mm Hg,bradypnea of less than 12/min, oxygen desaturation of less than 90%, seizures or a Glasgow Coma Scale score of less than 14)
* pregnancy
* drug addiction
* Patient who had already received a morphinic (within 6 hours) or anxiolitic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-05; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with pain relief (with a NRS score of 3/10 or lower) | 15 minutes after the first injection

SECONDARY OUTCOMES:
pain score comparisons | every 5 minutes within the first 30 minutes
pain and anxiety comparisons | 15 minutes after the first injection
comparison of adverse events | one hour after the first injection
patient and investigator satisfaction with analgesia | 30 minutes after the firest injection
assessment of post traumatic anxiety, stress and other related disorders | 2 days
assessment of post traumatic anxiety, stress and other related disorders | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis DUCASSE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Universty Hospital Toulouse SAMU 31, Toulouse, France